CLINICAL TRIAL: NCT00784251
Title: Validating PROMIS Instruments in Back and Leg Pain
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Dagmar Amtmann, Study Principal Investigator, University of Washington
Other Study IDs: 33606-J; 5U01AR052171-02 (NIH)
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Leg Pain; Back Pain
Keywords: Pain; Leg pain; Back pain; PROMIS
MeSH Terms: conditions — Back Pain; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Patient-Reported Outcomes Measurement Information System (PROMIS) is an NIH Roadmap initiative to develop a computerized system measuring patient-reported outcomes in respondents with a wide range of chronic diseases and demographic characteristics. In the first four years of its existence, the PROMIS network developed item banks for measuring patient-reported outcomes in the areas of pain, fatigue, emotional distress, physical function, and social functioning. During the item banking process, the PROMIS network conducted focus groups, individual cognitive interviews, and lexile (reading level) analyses to refine the meaning, clarity, and literacy demands of all items. The item banks were administered to over 20,000 respondents and calibrated using models based on item response theory (IRT). Using these IRT calibrations, computerized adaptive test (CAT) algorithms were developed and implemented. The network has designed a series of studies using clinical populations to evaluate the item attributes, examine their utility as CATs, and validate the item banks. More information on the PROMIS network can be found at www.nihpromis.org.

DETAILED DESCRIPTION:
The University of Washington Center on Outcomes Research in Rehabilitation (UWCORR) is a member of the Patient Reported Outcomes Information System (PROMIS) Network. PROMIS is funded by the NIH Roadmap initiative, working to improve the efficiency and accuracy of measuring patient-reported outcomes. UWCORR works collaboratively with five research sites (Stanford University, Duke University, State University of New York, University of Pittsburgh, and University of North Carolina) and a Statistical Coordinating Center (NorthShore University HealthSystem).

Collectively, the goal of the PROMIS Network is to create a publicly available system that can be periodically added to and modified and that allows clinical researchers to access a common repository of items and computerized adaptive tests. The first step in achieving this goal was to build item pools and develop core questionnaires that measure key health outcome domains that are manifested in a variety of disabilities and chronic conditions. The resulting six item banks cover the domains of pain, fatigue, social health, physical functioning, emotional functioning, and sleep-wake functioning.

The next step in this process is to validate the PROMIS item banks and to examine their utility as computerized adaptive tests (CATs) with individuals diagnosed with a variety of chronic conditions and disabilities. At UWCORR, we will recruit patients with back and leg pain who were treated with epidural steroid injections. This protocol is aimed at comparing the psychometric properties of the PROMIS item banks with non-PROMIS 'gold standard' instruments, diagnostic data, and medical records. We will compare de-identified data from this study with de-identified data from other PROMIS research centers.

ELIGIBILITY:
Inclusion Criteria:

* Back pain for at least 6 weeks
* Scheduled for any kind of spinal injection (i.e. epidural steroid injection, facet joint injection or sacroiliac joint injection) recommended by clinic physician

Exclusion Criteria:

* Not scheduled for ESI
* Has dementia or other cognitive impairments that would interfere with questionnaire completion
* Lumbar surgery within the last year; unstable neurological symptoms (e.g., experiencing bowel or bladder incontinence, numbness in groin area, new or worsening weakness in legs, or new numbness or tingling in legs); cauda equine syndrome; cancer; spinal cord injury (SCI); vertebral fractures; or multiple sclerosis (MS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with back and leg pain who are scheduled for epidural steroid injections and who have had pain for at least 6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
PROMIS measures

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar Amtmann, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Harborview Medical Center, Seattle, Washington
  - UWMC Sports and Spine Physicians, Seattle, Washington